CLINICAL TRIAL: NCT05765955
Title: A Randomized, Double-blind, Placebo-controlled, Multiple Ascending Dose Study to Evaluate Safety, PK and the Immunosuppressive Effects of p38 MAPK Inhibitor POLB 001 on the Intradermal and Intravenous LPS Challenge Response in Healthy Volunteers
Brief Title: Effects of p38 MAPK Inhibitor POLB 001 on in Vivo LPS Challenge Responses
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Poolbeg Pharma plc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CHDR2149
Record Dates: First submitted 2022-07-28; First posted 2023-03-13 (Actual); Last update posted 2023-03-14 (Actual); Status verified 2023-03

CONDITIONS: Influenza, Human
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- POLB 001 30 mg (Active Comparator)
  Interventions: Drug: POLB 001
- POLB 001 70 mg (Active Comparator)
  Interventions: Drug: POLB 001
- POLB 001 150 mg (Active Comparator)
  Interventions: Drug: POLB 001
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: POLB 001 — Investigational Medicinal Product
  Arms: POLB 001 150 mg; POLB 001 30 mg; POLB 001 70 mg
Drug: Placebo — Matching Placebo
  Arms: Placebo

SUMMARY:
A single center trial to evaluate the effect of POLB 001 on inflammatory responses following an intradermal LPS challenge in healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male volunteers aged 18 to 55 years, inclusive.
2. BMI in the range of 18 to 32 kg/m2 a minimum body weight of 50 kg.
3. Fitzpatrick skin type I-III.
4. Able to give written informed consent and willing to comply with all study-related procedures.
5. Has the ability to communicate well with the Investigator in the Dutch language and willing to comply with the study restrictions.

Exclusion Criteria:

1. (A history of) any clinically significant medical condition or abnormalities, as judged by the investigator.
2. History of sepsis, cardiovascular disease or malignancy.
3. History of trauma with likely damage to the spleen or surgery to spleen.
4. History of alcohol or drug abuse.
5. Any clinically significant febrile illness 30 days preceding study Day 1.
6. History of serious bleeding.
7. Clinical evidence of significant or unstable medical illness including neurological, hematological, cardiovascular (including clinically significant arrhythmia), hepatic, pulmonary, metabolic, gastrointestinal, renal, psychiatric, endocrine, or infectious diseases or malignancies. Subjects who have had splenectomy.
8. Previous participation in a systemic (i.v./inhaled) LPS challenge trial within a year before the first study day.
9. Have any current and / or recurrent pathologically, clinically significant skin condition at the lower forearms (i.e., atopic dermatitis) including tattoos.
10. Antibiotic use, operation or intervention by surgeon/dentist within one month before the first study day.
11. Subjects who have used any prescribed or non-prescribed systemic or topical medication (including herbal remedies) within 7 days of the first dose administration, or less than 5 half-lives (whichever is longer), and during the study (except for vitamin/mineral supplements) unless, in the opinion of the Investigator, the medication will not interfere with the study procedures or compromise safety.
12. Subjects who have received any medications, including St John's Wort, known to chronically alter drug absorption or elimination processes within 30 days of the first dose administration unless, in the opinion of the Investigator, the medication will not interfere with the study procedures or compromise safety.
13. Any active inflammatory or infectious disease (e.g., periodontitis).
14. Known immunodeficiency.
15. Positive test results for Hepatitis B, Hepatitis C, HIV antibody.
16. Subjects who consume on average more than 3 units of alcohol per day (one alcohol unit =1 beer [12 oz] =1 wine [5 oz] =1 spirits [1.5 oz]) or are unable to abstain from using alcohol during the study

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2022-07-22 (Actual); Primary Completion 2022-12-14 (Actual); Study Completion 2022-12-16 (Actual)

PRIMARY OUTCOMES:
Effect of intradermal LPS challenge | 16 days
  To evaluate the effect of POLB 001 on inflammatory responses following an intradermal LPS challenge in healthy volunteers
  Endpoints:
  Skin response by imaging
  - Erythema (multispectral imaging) (Clinician's Erythema Assessment (CEA) Scale)
Effect of intradermal LPS challenge | 16 days
  To evaluate the effect of POLB 001 on inflammatory responses following an intradermal LPS challenge in healthy volunteers
  Endpoints:
  Blister exudate analysis
  - Flow cytometry (neutrophils, monocyte subsets, T cells, B cells, NK cells, dendritic cells) (10*9/L)
Effect of intradermal LPS challenge | 16 days
  To evaluate the effect of POLB 001 on inflammatory responses following an intradermal LPS challenge in healthy volunteers
  Endpoints:
  Blister exudate analysis
  - Cytokines (IL-6, IL-8, TNF, IL-1β) (pg/mL)
Effect of intravenous LPS challenge | 16 days
  To evaluate the effect of POLB 001 on inflammatory responses following an intravenous LPS challenge in healthy volunteers
  Endpoints:
  Blood
  - Cytokines (IL-6, IL-8, IL-10, TNF, IL-1β) (pg/mL)

CONTACTS AND LOCATIONS:
Locations (1):
- Centre for Human Drug Research, Leiden, Netherlands

IPD SHARING:
Plan to Share IPD: No